CLINICAL TRIAL: NCT06335979
Title: A Phase Ib, Open-label, Ascending Dose Study With Step-up Doses to Assess Safety, Tolerability, and Pharmacokinetics of PIT565 in Participants With Systemic Lupus Erythematosus (SLE).
Brief Title: An Ascending Dose Study of PIT565 in Participants With Systemic Lupus Erythematosus (SLE).
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CPIT565B12101; 2023-510025-14-00 (Other: EU CT)
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus, SLE
Keywords: Systemic lupus erythematosus; SLE; ascending dose; B cells
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Cohort 1 (Experimental): Dose level 1
  Interventions: Drug: PIT565
- Cohort 2 (Experimental): Dose level 2
  Interventions: Drug: PIT565
- Cohort 3 (Experimental): Dose level 3
  Interventions: Drug: PIT565
- Cohort 4 (Experimental): Dose level 4
  Interventions: Drug: PIT565
- Cohort 5 (Experimental): Dose level 5
  Interventions: Drug: PIT565
- Cohort 6 (Experimental): Dose level 6
  Interventions: Drug: PIT565
- Cohort 7 (Experimental): Dose level 7
  Interventions: Drug: PIT565
- Cohort 8 (Experimental): Dose level 8
  Interventions: Drug: PIT565

INTERVENTIONS:
Drug: PIT565 — In each cohort, there will be 3 sentinel participants. Additional participants might be added depending on safety and observed biological activity.

SUMMARY:
The purpose of the study is to determine the safety, tolerability, and pharmacokinetics of PIT565 in participants with SLE

DETAILED DESCRIPTION:
This is an open-label, ascending dose, uncontrolled study in participants with SLE systemic lupus erythematosus (SLE). PIT565 will be administered subcutaneously (s.c.) following premedication.

Up to 8 cohorts are planned. Every cohort will have 3 sentinel participants and, depending on safety as well as observed biological activity, may have up to 3 additional optional participants (up to 6 participants per cohort). The decision to escalate the dose from one cohort to the next will be based both on safety and PD data. After the identification of a dose level that has been declared safe and has induced predefined B cell depletion in 100% of the participants (candidate dose level), the cohort from this candidate dose level can optionally be enriched with 6 additional participants (up to a total of 12 participants).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE according to the 2019 ACR/EULAR criteria
* Documentation of SLE autoantibodies
* Active SLE disease, as demonstrated by a SLEDAI-2K ≥ 4 at screening
* Failure to respond to standard-of-care medicines for the treatment of SLE as detailed in the protocol
* Immunization against pneumococcus, meningococcus, influenza, and COVID-19

Exclusion Criteria:

* Severe SLE-related organ damage dysfunction or life-threatening disease at screening.
* Any acute, severe lupus-related flare during screening that needs immediate treatment such as acute CNS lupus (e.g., psychosis, epilepsy) or catastrophic antiphospholipid syndrome.
* Presence of severe lupus kidney disease as defined by worsening proteinuria or estimated glomerular filtration rate (eGFR) which in the opinion of the Investigator requires immunosuppressive induction or maintenance treatment at screening.
* History or current diagnosis of ECG or cardiac abnormalities indicating a significant risk of safety for participants.
* Use of prohibited medication defined in the protocol.
* Clinically significant active, opportunistic, chronic or recurrent infection (including, HIV, HBV, HCV) confirmed one month prior to or during screening.
* Serious medical illness likely to interfere with participation in this clinical study.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant from menarche until becoming post-menopausal, unless they are using highly effective methods of contraception

Other protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2027-07-09 (Estimated); Study Completion 2027-07-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse events (AEs) and Serious Adverse events (SAEs) | From Study Day 1 until Study Day 180
  Safety assessments of PIT565 including changes in vital signs, electrocardiograms (ECG) and laboratory results from baseline

SECONDARY OUTCOMES:
Maximum Observed Blood Concentrations (Cmax) | From pre-dose Day 1 until Day 29
  Cmax is the maximum (peak) observed plasma, blood, serum, or other body fluid drug concentration after single dose administration (mass x volume-1).
Presence/absence of Anti-drug Antibodies | From pre-dose Day 1 until Day 180
  Assess immunogenicity of PIT565 at pre-dose, and over time

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- Novartis Investigative Site, Sofia, Bulgaria
- Novartis Investigative Site, Beijing, China
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Mainz
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
- Novartis Investigative Site, Leiden, South Holland, Netherlands
- Spain (2):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, Barcelona
- Switzerland (2):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No